CLINICAL TRIAL: NCT07345247
Title: RAdiation SEgmentectomy With REsin Microspheres (RASEREM) Study
Acronym: RASEREM
Status: Recruiting | Type: Observational
Sponsor: Ankara University (Other)
Collaborators: Sirtex Medical (Industry)
Responsible Party: Principal Investigator, Cigdem Soydal, Prof, Ankara University
Other Study IDs: RASEREM
Record Dates: First submitted 2025-12-28; First posted 2026-01-15 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Liver Cancer, Adult
Keywords: Liver Cancer; Radioembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Radiation Segmentectomy Group: Patients who will receive radioembolization for radiation segmentectomy intent

SUMMARY:
Radiation segmentectomy (RS) refers to selective infusion of Y-90 microspheres to the tumor bearing hepatic segment of hepatic artery. Majority of the data on RS is based on the Glass microspheres experience. Due to different properties of Resin and Glass microspheres description of dose limits to the segment for effectiveness of treatments with Resin microspheres are needed.

Based on this background in this study it is aimed to evaluate the safety and efficacy of RS with resin microspheres in HCC patients. Secondly, it is planned to describe the dose limits for complete radiological response.

DETAILED DESCRIPTION:
Radiation segmentectomy (RS) refers to selective infusion of Y-90 microspheres to the tumor bearing hepatic segment of hepatic artery. It was first described in 2011 and has been demonstrated to be a safe and reliable therapy able to deliver a curative intent high dose of selective ablative radiation for the treatment of hepatocellular carcinoma (HCC). This approach is gained to the radioembolization to a notable position in today's established algorithm for the multidisciplinary management of HCCs. Majority of the data on RS is based on the Glass microspheres experience. Due to different properties of Resin and Glass microspheres description of dose limits to the segment for effectiveness of treatments with Resin microspheres are needed.

In a recent retrospective study it is demonstrated that RS with resin microspheres are safe and effective In comparison to glass microspheres evet with lower radiation doses to the tumor. Despite this data on the effectiveness and safety of RS with resin microspheres in the multidisciplinary meeting I noticed that nuclear medicine specialist and interventional radiologist form our country rely on the use glass microspheres in the RS setting. As a nuclear medicine specialist who perform RS with resin microspheres I need to show the success of resin microspheres in RS with a multicenter prospective study. I believe that this multicenter experience would change clinical practice in our country and the scientific data that we will have would place the resin microspheres to its real place in the RS setting worldwide.

Based on this background in this study it is aimed to evaluate the safety and efficacy of RS with resin microspheres in HCC patients. Secondly, it is planned to describe the dose limits for complete radiological response.

All post treatment Y-90 PET images will be used for dosimetric estimations. Single compartment dosimetry will be performed in the treating center. If the center do not have dosimetric software calculation will be performed by PI in the Ankara University by using Slicer 3D software and a dedicated module for liver dosimetry. Response to the treatment will be evaluated by MRI imaging with liver specific contrast agent after 3 and 6 months treatment. mRECIST criteria will be used for evaluation. Additionally, change in serum tumor markers levels will be evaluated. Standard clinical protocol included clinical and laboratory evaluation at baseline, two weeks, one month, and three months after treatment. Laboratory markers for analysis will be: serum albumin, total bilirubin, alkaline phosphatase (AP), gamma-glutamyltransferase (GGT), aspartate aminotransferase (AST), and alanine transaminase (ALT). All events will be evaluated using the Common Terminology Criteria for Adverse Events (CTCAE) version 5. Preexisting toxicities will be excluded unless they exacerbated after treatment.

Totally 150 patients are planning to include the analysis. ROC analysis will be use for determination of optimal cutoffs for mean tumor and segment absorbed doses to predict response and complete response. Multivariate regression model will be used for analysis of multiple factors for response. Lineer regression model will be perform for whole liver absorbed dose and toxicity evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years
* Underwent RE as a RS intent (have single or <3 tumors in same or neighboring 2 segments) for the treatment of HCC or metastatic tumor to liver.
* Presence of extrahepatic disease
* Tumor size less than 8 cm
* Child Pugh Score <B9

Exclusion Criteria:

* Presence of macrovascular invasion,
* Presence of extrahepatic disease,
* Cholangiocarcinoma or mixed HCC-cholangiocarcinoma
* Not willing to attend follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will include the patients who will receive radioembolization for radiation segmentectomy intent for primary or secondary liver tumors
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of radiation segmentectomy | 3 months after treatment
  Evaluation of response with modified RECIST criteria

SECONDARY OUTCOMES:
Safety of radioembolization in radiation segmentectomy intent | 3 months after treatment
  Evaluation of toxicity of radiation segmentectomy at the 3 month of treatment with CTCAE grading

CONTACTS AND LOCATIONS:
Locations (20):
- Turkey (Türkiye) (20):
  - Acibadem Adana Hospital, Adana
  - Adana City Hospital, Adana
  - Cukurova University, Adana
  - Bilkent City Hospital, Ankara
  - Gulhane Education and Research Hospital, Ankara
  - Hacettepe University, Ankara
  - Pamukkale University, Denizli
  - Gazi Yasargil Education and Research Hospital, Diyarbakır
  - Cam ve Sakura Education and Reseach Hospital, Istanbul
  - Istanbul Unicersity Cerrahpasa Medical School, Istanbul
  - Istanbul University Capa Medical School, Istanbul
  - Marmara University, Istanbul
  - Acibadem Izmir Hospital, Izmir
  - Ege University, Izmir
  - Katip Celebi Education and Research Hospital, Izmir
  - Erciyes University, Kayseri
  - Kocaeli University, Kocaeli
  - Konya Selcuk University, Konya
  - Inonu University, Malatya
  - Mersin City Hospital, Mersin

IPD SHARING:
Plan to Share IPD: Undecided